CLINICAL TRIAL: NCT01911403
Title: Efficacy Superiority of Angio-Seal™ vs. Manual Compression in Interventional Radiology
Brief Title: AGIR Study: Angio-Seal in Interventional Radiology
Acronym: AGIR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment rate.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV08025POVC
Record Dates: First submitted 2011-04-14; First posted 2013-07-30 (Estimated); Results first posted 2015-03-11 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Vascular Access Complication
Keywords: Femoral Artery puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Angio-Seal (Active Comparator): Closure procedure by Angio-Seal
  Interventions: Device: Angio-Seal
- Manual compression (Active Comparator): Closure procedure by manual compression
  Interventions: Procedure: Manual compression

INTERVENTIONS:
Procedure: Manual compression — Closure procedure by Manual compression
  Arms: Manual compression
Device: Angio-Seal — Closure procedure by angio-Seal
  Arms: Angio-Seal

SUMMARY:
Clinical study in patients undergoing any intervention requiring vascular access to the femoral artery. The study compares Angio-Seal™ vs. Manual Compression with regard to control the vascular access.

It is designed to demonstrate superiority of the Angio-Seal™ with an unchanged risk-profile.

DETAILED DESCRIPTION:
Patients will have their puncture closure randomly performed by one of these approved methods: Angio-Seal™ Closure device or Manual Compression.

Patients will be enrolled in the study during 12 months, with a follow-up period of 2 weeks (± 1 week).

The randomization will be stratified according to the type of procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years Interventional Radiology procedures with Femoral Artery puncture (4 French - 8 French Introducers)
* Patient available for follow-up at 2 weeks
* Patients who are willing to participate and have signed an Ethic Committee approved patient informed consent.

Exclusion Criteria:

* Access unsuitable for use of Angio-Sea
* Presence of calcification at the puncture site
* Presence of visible hematoma at the end of the procedure
* Patients who are unable to comply with the follow-up schedule based on their geographic location or for any reason.
* Patients who are pregnant.
* Patients currently participating in a clinical investigation that includes an active treatment arm.
* Contraindication for ambulation at 2 hours after the end of the procedure
* Patients with a life expectancy of less then 1 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2010-12; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Alberto Mingo, PhD., Principal Investigator — Hospital Universitario de La Princesa, Madrid; Dr. Paolo Morgado, PhD., Principal Investigator — Hospital de São João, E.P.E.
Locations (2):
- Hospital de São João, E.P.E., Porto, Portugal
- Hospital Universitario de La Princesa, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Angio-Seal | Manual Compression
Started | 61 | 62
Completed | 52 | 59
Not Completed | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Angio-Seal | Manual Compression | Total
Number analyzed (Participants) | 61 | 62 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.77 (15.15) | 60.92 (13.55) | 60.84 (14.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 39
  Male | 39 | 45 | 84

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Mobilization Time Between 0-4 Hours
Description: Mobilization Time is the time that patient gets the authorization to flex the leg, sit or walk.
Time Frame: At discharge
Measure: Number; unit: participants
Arm/Group | Angio-Seal | Manual Compression
Number analyzed (Participants) | 61 | 62
participants | 52 | 14

2. Secondary Outcome: Number of Patients With Mobilization Time Between 4-48 Hours
Description: Mobilization Time is the time that patient gets the authorization to flex the leg, sit or walk.
Time Frame: At discharge
Measure: Number; unit: participants
Arm/Group | Angio-Seal | Manual Compression
Number analyzed (Participants) | 61 | 62
participants | 9 | 48

3. Secondary Outcome: Number of Patients With Any Complications
Description: Number of patients with any complications since the puncture closure until 2 weeks ± 1 week.
  The complications are related to the puncture closure evaluated at closure, discharge and follow-up. These include hematoma, Inferior limb ischemia, prolonged pain at puncture site, puncture site local infection, pseudoaneurysm, significant bleeding and vessel occlusion.
Time Frame: At puncture closure procedure, at discharge and at follow up (2 weeks+/-1 week)
Measure: Number; unit: participants
Arm/Group | Angio-Seal | Manual Compression
Number analyzed (Participants) | 61 | 62
participants | 6 | 6

4. Secondary Outcome: Number of Patients With Time to Hemostasis Between 0-4 Minutes
Description: Time to hemostasis is the time from the beginning of closure procedure, until the physician take away their hands from the patient, regardless the closure procedure, and confirm the "stop of bleeding".
Time Frame: At puncture closure
Measure: Number; unit: participants
Arm/Group | Angio-Seal | Manual Compression
Number analyzed (Participants) | 61 | 62
participants | 54 | 1

5. Secondary Outcome: Number of Patients With Time to Hemostasis Between 4-60 Minutes
Description: as for outcome 4
Time Frame: At puncture closure
Measure: Number; unit: participants
Arm/Group | Angio-Seal | Manual Compression
Number analyzed (Participants) | 61 | 62
participants | 7 | 60

6. Secondary Outcome: Time to Discharge From Interventional Radiology Department
Description: Time that the physician grants the patient the discharge order from the Radiology Department. If the patients has order to be hospitalized up to 24h after the puncture closure by the radiologist, then, the discharge from the radiology department will be 24h, even if the patient needs to continue hospitalized in other department.
Time Frame: At discharge
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Angio-Seal | Manual Compression
Number analyzed (Participants) | 61 | 62
hours | 3.70 (7.79) | 3.64 (9.61)

7. Secondary Outcome: Percentage of Patients With Angio-Seal™ Deployment Success
Description: According the physician criteria, it will be "YES" If the anchor was deliver properly, the absorbable component remain in the correct point of the arterial puncture and no bleeding in the skin puncture.
Time Frame: At puncture closure
Population: Only patients in the Angio-Seal arm is analyzed
Measure: Number; unit: percentage of patients
Arm/Group | Angio-Seal
Number analyzed (Participants) | 61
percentage of patients | 95.1

ADVERSE EVENTS:
Time Frame: 2 weeks (+/- 1 week)
Arm/Group | Angio-Seal | Manual Compression
Serious Adverse Events (participants affected / at risk) | 3/61 | 6/62
Other Adverse Events (participants affected / at risk) | 7/61 | 2/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Angio-Seal (N=61) | Manual Compression (N=62)
Deterioration of general condition (General disorders) | 0 (0) | 1 (1) — DETERIORATION OF THE GENERAL CONDITION OF THIS GERIATRIC PATIENT
Bleeding (Surgical and medical procedures) | 0 (0) | 1 (1) — BLEEDING OF THE PUNCTURE SITE
Superficial Perforation femoral artery (Surgical and medical procedures) | 0 (0) | 1 (1) — PERFORATION SUPERFICIAL FEMORAL ARTERY
Significant bleeding (Surgical and medical procedures) | 0 (0) | 1 (1) — SIGNIFICANT BLEEDING AFTER MANUAL COMPRESSION WITH PROLONGATION OF MANUAL COMPRESSION AND PROLONGED HOSPITAL STAY.
Hematoma (Surgical and medical procedures) | 1 (1) | 0 (0) — HEMATOMA AFTER 24 HOURS AT PUNCTURE SITE
Hepatic Abcess (Hepatobiliary disorders) | 0 (0) | 1 (1) — HEPATIC ABSCESS. DISCHARGE ON 3/06/2011
Edematoascitis (General disorders) | 0 (0) | 1 (1) — FEVER, EDEMATOASCITIS DECOMPENSATIS, INFERIOR EXTREMITIES CELLULITIS GREATER IN COUNTER LATERAL PUNCTION SITE
Minor Stroke (Cardiac disorders) | 1 (1) | 0 (0) — MINOR STROKE LEFT SIDE
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1) — SERIOUS URINARY TRACT INFECTION IN AN ELDERLY PERSON
Vessel stenosis (Surgical and medical procedures) | 1 (1) | 0 (0) — PROLONGED PAIN AT THE PUNCTURE SITE. VESSEL STENOSIS
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Angio-Seal (N=61) | Manual Compression (N=62)
Hematoma (Surgical and medical procedures) | 0 (0) | 1 (1) — BIGGER BRUISE : SMALL HEMATOMA LESS THAN 6 CM SIGNALED BY THE PATIENT
Bleeding (Surgical and medical procedures) | 1 (1) | 0 (0) — FAILURE OF INTRODUCTION OF THE INTRODUCER OF THE ANGIO-SEAL WITH SIGNIFICANT BLEEDING.
Bruise (Surgical and medical procedures) | 1 (1) | 0 (0) — BIGGER BRUISE OF THE PUNCTURE AREA AND WENT TO A GENERAL PRACTITIONER
Headache and vomits (Vascular disorders) | 1 (1) | 0 (0) — ACUTE HEADACHE + ONE TIME VOMITING AFTER CAROTID STENTING
Hematoma (Surgical and medical procedures) | 0 (0) | 1 (1) — HEMATOMA AFTER 5 DAYS OF INTERVENTIONAL PROCEDURE
Bruise (Surgical and medical procedures) | 1 (1) | 0 (0) — BRUISE IN THE PUNCTION AREA STILL PRESENT AT PHONE CALL VISIT
Bleeding (Surgical and medical procedures) | 1 (1) | 0 (0) — BLEEDING AFTER CLOSURE PROCEDURE
Bleeding (Surgical and medical procedures) | 1 (1) | 0 (0) — BLEEDING AFTER CLOTURE PROCEDURE
Pain (Surgical and medical procedures) | 1 (1) | 0 (0) — SLIGHT PAIN AT PUNCTURE SITE
Hematoma (Surgical and medical procedures) | 1 (1) | 0 (0) — HEMATOMA DURING THE PROCEDURE RELATED TO CALCIFICATION
Hematoma (Surgical and medical procedures) | 1 (1) | 0 (0) — SMALL HAEMATOMA (+/- 1 CM)
Pain (Surgical and medical procedures) | 1 (1) | 0 (0) — PAIN IN THE PUNCTURE AREA

LIMITATIONS AND CAVEATS:
This study has been early terminated on 15 May 2014 due to low enrollment rate and the publication of other larger studies about closure device versus manual compression.This lead to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other